CLINICAL TRIAL: NCT05906446
Title: Feasibility of a Multicomponent Frailty Intervention During Post-acute Rehabilitation in Skilled Nursing Facilities
Brief Title: Post-acute Multicomponent Frailty Intervention
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Sandra Shi, Instructor of Medicine, Hebrew SeniorLife
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00068129
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Regular exercise sessions incorporating balance, resistance training, and walking to accommodate diminished endurance, with synergistic protein and nutritional supplementation
  Interventions: Other: Multicomponent (Exercise + Protein Supplementation)

INTERVENTIONS:
Other: Multicomponent (Exercise + Protein Supplementation) — * Exercises selected from a pre-specified list, reassessed weekly
  * Participants will receive individualized exercise sessions, (e.g. 15-30 minutes per session, one session per day, offered five times a week)
  * Participants will also be offered a protein supplement within 30 min of exercise.
  * Sessions will be supervised

SUMMARY:
The goal is to test feasibility of a frailty intervention, including exercises and nutritional supplementation.

DETAILED DESCRIPTION:
The frailty intervention includes frequent short exercise sessions incorporating balance, resistance training, and walking to accommodate diminished endurance, with synergistic protein and nutritional supplementation, delivered on top of usual care in the post-acute Skilled Nursing Facility (SNF) setting. There is no control group.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling before hospitalization
* Age ≥ 65 years
* Admitted to SNF directly from inpatient hospitalization
* English speaking
* Mild Frailty or worse, as measured by a Clinical Frailty Scale

Exclusion Criteria:

* Discharged from Emergency Department
* Non-community discharge plan on admission (e.g. plan to discharge to hospice)
* Nothing per oral (NPO) dietary status
* Presence of any feeding tube
* Chronic kidney disease stage IV or worse
* Clinician refusal
* Inability or refusal to consume intervention products (e.g. allergies to protein supplement)
* Inability to consent to study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Estimated average <1 month
  Feasibility will be determined by assessing 1) the proportion of eligible patients enrolled, and 2) the proportion of participants adherent to the intervention
  Range: 0-100% (higher values indicate higher feasibility).

SECONDARY OUTCOMES:
Gait Speed | Discharge (on average between 2-3 weeks)
  Walking speed measured in m/s
Grip Strength | Discharge (on average at 2-3 weeks)
  Dominant Hand Grip Strength measured in Kg (higher values indicate better performance)
The Patient Reported Outcomes Measurement Information System (PROMIS Global Health v1.2) | Discharge (on average at 2-3 weeks)
  The PROMIS Scale v1.2 - Global Health (also referred to as PROMIS-10) is a ten-item patient reported measure of physical, mental and social health. Items query general health, quality of life, physical health, mental health, satisfaction with discretionary social activities, carrying out every day physical activities, pain, fatigue, satisfaction with social roles, and emotional problems (Hays et al., 2009).
  Physical Health (physical health, physical function, pain, and fatigue items) and Mental Health (quality of life, mental health, satisfaction with discretionary social activities, and emotional problem items) (Hays et al., 2009).
  T scores for both Physical and Mental Health scales.
Modified Barthel Index | Discharge (on average at 2-3 weeks)
  Assessment of functional disability based on 10 activities of daily life (ADLs). Range 0-10 with high values indicating better performance.
Adherence to exercise | Entire study period (on average over 2-3 weeks)
  Proportion of sessions with exercise during the intervention period
  Range: 0-100% (higher values indicate better adherence)
Adherence to supplementation | Entire study period (on average over 2-3 weeks)
  Proportion of oral nutritional supplement consumed over the total number of supplements during the intervention period per self-report
  Range: 0-100% (higher values indicate better adherence)

OTHER OUTCOMES:
Length of stay | Entire study period (on average over 2-3 weeks)
  Length of admission to SNF
Hospital readmission | Entire study period (on average over 2-3 weeks)
  Proportion of participants who are readmitted to the hospital during SNF stay
Community Discharge | Entire study period (on average over 2-3 weeks)
  Proportion of participants who are discharged to the community from SNF stay
Falls | Entire study period (on average over 2-3 weeks)
  Proportion of participants who experience a fall, as documented in the medical record, during SNF stay

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Shi, MD MPH, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No